CLINICAL TRIAL: NCT01657994
Title: Combined Functional Electrical Stimulation & Robotic Gait Training for Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Cerebral Palsy International Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-796-10
Record Dates: First submitted 2012-05-17; First posted 2012-08-06 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; gait training; robotic; functional electrical stimulation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- therapy plus fes (Experimental): robotic gait training plus functional electrical stimulation
  Interventions: Other: Combined functional electrical stimulation and robotic gait training

INTERVENTIONS:
Other: Combined functional electrical stimulation and robotic gait training — up to 18 sessions of approximately 45 minutes occurring over up to 9 weeks
  Other Names: Lokomat; RT-50

SUMMARY:
The purpose of this research study is to learn more about the usefulness of a physical therapy treatment that combines robot-assisted walking with electrical impulses that help to make muscles contract. This treatment is intended for children with cerebral palsy. Up to eleven children with cerebral palsy will receive up to 18 treatments and will have several evaluations before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* GMFCS II, III, or IV cerebral palsy
* 5-12 years of age
* meet safety criteria for robotic gait training (<300 lbs, intact skin, femoral length 21-47 cm, ability to follow simple instructions)
* meet safety criteria for functional electrical stimulation (voluntary hip and knee muscle contraction, intact skin)

Exclusion Criteria:

* planned major intervention during study period
* contractures that interfere with upright stance
* history of non-traumatic long bone fracture or clinically significant osteoporosis
* significant concurrent illness
* significant condition not typically associated with cerebral palsy

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in Gross Motor Function Measure-66 using multiple baseline assessments | 4 times (9-0 weeks) before treatment, 3 times (6-12 weeks) after treatment

SECONDARY OUTCOMES:
Change in strength via myometry | 4 times (9-0 weeks) before treatment, 3 times (6-12 weeks) after treatment
Change in Observational Gait Scale | 4 times (9-0 weeks) before treatment, 3 times (6-12 weeks) after treatment
Change in Modified Ashworth Scale | 4 times (9-0 weeks) before treatment, 3 times (6-12 weeks) after treatment
Change in Goniometry at the knee | 4 times (9-0 weeks) before treatment, 3 times (6-12 weeks) after treatment
Change in 6 minute walk | 4 times (9-0 weeks) before treatment, 3 times (6-12 weeks) after treatment
Change in 10 meter walk | 4 times (9-0 weeks) before treatment, 3 times (6-12 weeks) after treatment
Change in Children's Assessment of Participation and Enjoyment | 4 times (9-0 weeks) before treatment, 3 times (6-12 weeks) after treatment
Change in Cerebral Palsy Quality of Life Questionnaire | 4 times (9-0 weeks) before treatment, 3 times (6-12 weeks) after treatment
Change in Canadian Occupational Performance Measure | 4 times (9-0 weeks) before treatment, 3 times (6-12 weeks) after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jilda Vargus-Adams, MD MSc, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States